CLINICAL TRIAL: NCT02537392
Title: Primary Prevention of Multi-micronutrient Supplementation During Peri-conception Against Congenital Heart Disease: A Community-based Randomised Controlled Trial in China
Brief Title: Multi-micronutrient Supplementation During Peri-conception and Congenital Heart Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xi'an Jiaotong University (Other)
Responsible Party: Principal Investigator, Jiaomei Yang, PhD candidate, Xi'an Jiaotong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NSFC81230016
Record Dates: First submitted 2015-08-27; First posted 2015-09-01 (Estimated); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Vitamin B Complex; Folic Acid; Iron

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Vitamin B Complex and Folic Acid (Experimental): Daily supplements containing vitamin B1 (2 mg), vitamin B2 (2 mg), vitamin B6 (2 mg), vitamin B12 (2 μg), calcium pantothenate (2 mg), nicotinamide (15 mg) and folic acid (0.4 mg).
  Interventions: Dietary Supplement: Vitamin B Complex and Folic Acid
- Iron and Folic Acid (Experimental): Daily supplements of iron (60 mg) and folic acid (0.4 mg).
  Interventions: Dietary Supplement: Iron and Folic Acid
- Folic Acid (Active Comparator): Daily supplement of 0.4 mg folic acid.
  Interventions: Dietary Supplement: Folic Acid

INTERVENTIONS:
Dietary Supplement: Vitamin B Complex and Folic Acid — Daily oral dose containing 2 mg vitamin B1, 2 mg vitamin B2, 2 mg vitamin B6, 2 μg vitamin B12, 2 mg calcium pantothenate, 15 mg nicotinamide and 0.4 mg folic acid.
  Arms: Vitamin B Complex and Folic Acid
Dietary Supplement: Iron and Folic Acid — Daily oral dose of 60 mg iron and 0.4 mg folic acid.
  Arms: Iron and Folic Acid
Dietary Supplement: Folic Acid — Daily oral dose of 0.4 mg folic acid.
  Arms: Folic Acid

SUMMARY:
The purpose of this study is to determine whether daily oral supplements of vitamin B complex along with folic acid or supplements of iron plus folic acid given to women during peri-conception can reduce the risk of congenital heart disease when compared with folic acid alone.

DETAILED DESCRIPTION:
Congenital heart disease (CHD) is among the most prevalent congenital abnormalities with an incidence of about 8-12/1,000 live births, and is also the leading cause of infant morbidity and death from birth defects. A series of studies pointed out that the poor nutritional status of the mother during peri-conception might be the important cause of CHD. In maternal folic acid/ vitamin B deficiency homocysteine accumulates in the serum, and elevated circulating homocysteine concentrations have been associated with the risk of CHD. However, it is still questionable whether multiple vitamin B supplements during peri-conception can reduce CHD risk more effectively compared with the supplement of folic acid alone. Moreover, one randomized controlled trial performed in Shaanxi China confirmed that the supplement of iron and folic acid during pregnancy can significantly reduce early neonatal deaths. It is noteworthy that one-fourth of newborn deaths are attributable to birth defects. Thus, it is worthwhile to investigate whether iron supplement can reduce the risk of CHD.

This community-based randomized controlled trial will assess and compare the impact of daily oral supplements of vitamin B complex along with folic acid or supplements of iron plus folic acid vs. folic acid alone given to women during peri-conception on CHD. It will also assess the effects of the three different supplementations on other pregnancy outcomes and maternal health. The study will be conducted in three rural poor counties including Xunyi, Changwu, and Bin, which are located in Shaanxi Province of Northwest China. All participants will sign informed consent before the study. The investigators hypothesize that the newborn infants of women receiving supplements of vitamin B complex along with folic acid or supplements of iron plus folic acid will experience a reduction in the prevalence of infants with the pulse oxygen saturation less than 95% and other adverse pregnancy outcomes compared with those receiving folic acid alone. The results of this trial will provide evidence needed to formulate policy on maternal micronutrient supplementation during peri-conception and the rationale for the necessary investment of public funds to implement appropriate programs against birth defects.

ELIGIBILITY:
Inclusion Criteria:

1. Women of reproductive age (15-49 years) who reside in the study areas;
2. Women who are prepared for pregnancy in 1-3 months or have already been pregnant for less than 20 months;
3. Women who have provided written informed consent.

Exclusion Criteria:

1. Women who have already taken supplements containing vitamin B complex, iron, or folic acid for more than two weeks at enrollment;
2. Women who have given birth to children with congenital heart disease or other birth defects before;
3. Women with diabetes;
4. women with severe heart, liver or kidney disease.

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7315 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Neonatal pulse oximetry oxygen saturation measured by pulse oximetry | 6-72 hours after delivery
  Neonatal pulse oximetry oxygen saturation (SpO2) is tested by pulse oximetry in babies aged between 6 h and 72 h after birth. Pulse oximetry testing is repeated 4 h later if the first measurement is between 90% and 95%. The result of SpO2 will be reported as a dichotomous variable, in which the result is deemed positive if an SpO2 less than 95% is obtained both on the right hand and on either foot on two measures, separated by 4 h; a difference between the two extremities was more than 3% on two measures, separated by 4 h; or any measure is less than 90%. The result of SpO2 will also be reported as a continuous variable.

SECONDARY OUTCOMES:
Incidence of congenital heart disease and the subtypes | Half a year after delivery
  Congenital heart disease will be diagnosed by trained clinicians with the help of echocardiography, pulse oximetry, clinical examination, cardiac surgery, or autopsy. The incidence of congenital heart disease and the subtypes will be reported in each group.
Incidence of birth defects and the subtypes | Half a year after delivery
  Birth defects will be diagnosed by trained clinicians. The incidence of birth defects and the subtypes will be reported in each group.
Birth weight measured by baby scale | Within 1 hours of delivery
  Birth weight will be measured within 1 hour of delivery using a baby scale with the precision to the nearest 50 gram.
Incidence of low birth weight | Within 1 hour of delivery
  Birth weight will be measured within 1 hour of delivery using a baby scale. The incidence of low birth weight will be reported in each group based on the criteria of birth weight less than 2500 gram.
Gestational age at birth | At delivery
  Gestational age at birth will be measured as completed days based on the last menstrual period.
Incidence of preterm birth | At delivery
  Gestational age at birth will be measured as completed days based on the last menstrual period. The incidence of preterm birth (infant born less than 37 weeks gestational age) will be reported in each group.
Incidence of perinatal mortality | Between 28 weeks of gestational duration and 7 days after delivery
  The incidence of perinatal mortality (Infants death between 28 weeks of gestational duration and 7 days after delivery) will be reported in each group.
Incidence of stillbirth | At delivery
  The incidence of stillbirth (infants death at delivery) will be reported in each group.
Incidence of neonatal mortality | First 28 days after birth
  The incidence of neonatal mortality (infants death during the first 28 days after birth) will be reported in each group.
Incidence of early neonatal mortality | First 7 days after birth
  The incidence of early neonatal mortality (infants death during the first 7 days after birth) will be reported in each group.
Incidence of pregnancy complications: hypertension, preeclampsia, antepartum haemorrhage, and infections | After enrollment until at delivery
  Pregnancy complications (hypertension, preeclampsia, antepartum haemorrhage, and infections) will be diagnosed by trained clinicians during antenatal care checks. All information will be recorded in the pregnant women's medical records of antenatal care checks and delivery. The incidence of hypertension, preeclampsia, antepartum haemorrhage, and infections among participants will be reported in each group.

CONTACTS AND LOCATIONS:
Overall Officials: Hong Yan, Professor, Principal Investigator — Xi'an Jiaotong University
Locations (1):
- Xi'an Jiaotong University College of Medicine, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mi B, Wen X, Li S, Liu D, Lei F, Liu R, Shen Y, Chen Y, Zeng L, Liu X, Dang S, Yan H. Vegetable dietary pattern associated with low risk of preeclampsia possibly through reducing proteinuria. Pregnancy Hypertens. 2019 Apr;16:131-138. doi: 10.1016/j.preghy.2019.04.001. Epub 2019 Apr 8. PMID 31056148